CLINICAL TRIAL: NCT01922466
Title: Clinical Research on the Efficacy and Safety of East-West Collaborative Treatment Using NSAIDs and BV on Chronic Cervical Pain; A Randomized, Controlled, Parallel, Pilot Study
Brief Title: East-West Collaboration Treatment Using Bee Venom Acupuncture and NSAIDs for Chronic Cervicalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Kyunghee University (Other); Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, Byung-Kwan Seo, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2012-019
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Non-specific, Uncomplicated Neck Pain
Keywords: chronic neck pain; combined treatment between conventional and complementary alternative medical treatment; bee venom acupuncture; NSAIDs
MeSH Terms: interventions — loxoprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bee Venom Acupuncture (Experimental)
  Interventions: Procedure: Bee Venom Acupuncture
- Loxoprofen (Experimental)
  Interventions: Drug: Loxoprofen
- EWCT : Bee Venom Acupucture and Loxoprofen (Experimental)
  Interventions: Procedure: Bee Venom Acupuncture; Drug: Loxoprofen

INTERVENTIONS:
Procedure: Bee Venom Acupuncture — Bee Venom 1:20,000 under BVA Increment Protocol
  - Increment Protocol as
  * 1st week - SC 0.2cc/day, 2 days/week
  * 2nd week - SC 0.4cc/day, 2 days/week
  * 3nd week - SC 0.8cc/day, 2 days/week
  Other Names: pharmacopuncture
  Arms: Bee Venom Acupuncture; EWCT : Bee Venom Acupucture and Loxoprofen
Drug: Loxoprofen — 60 mg/Tab, pers os 1Tab tid, for 3 weeks
  Other Names: Loxonin
  Arms: EWCT : Bee Venom Acupucture and Loxoprofen; Loxoprofen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of east-west collaborative treatment using bee venom acupuncture and NSAIDs on pain intensity, functional status and quality of life of patients with chronic cervicalgia

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* nonspecific, uncomplicated, chronic neck pain over 3 months
* volunteer can read and write in Korean, providing written informed consent

Exclusion Criteria:

* exhibited abnormalities on neurological examination
* radicular pain
* serious spinal disorders including malignancy, vertebral fracture, spinal infection or inflammatory spondylitis
* other chronic diseases that could affect or interfere with the therapeutic outcomes including cardiovascular disease, diabetic neuropathy, active hepatitis, fibromyalgia, rheumatoid arthritis, dementia or epilepsy
* previous spinal surgery or scheduled procedures during the study
* painful conditions induced by traffic accidents
* a substantial musculoskeletal problem generating pain from an area other than the neck
* conditions for which administration of BVA might not be safe including clotting disorders, administration of an anticoagulant agent, pregnancy and seizure disorders
* a documented hypersensitive reaction to previous BVA treatments, bee stings or insect bites
* positive reaction observed during a skin hypersensitivity test
* severe psychiatric or psychological disorders
* current use of corticosteroids, narcotics, muscle relaxants or herbal medicines to treat neck pain or any medication considered inappropriate by the investigator
* pending lawsuits or receipt of compensation due to neck pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for bothersomeness | Changes from baseline in VAS at 1st, 2nd, 3rd, 4th and 8th week follow-up

SECONDARY OUTCOMES:
Neck Disability Index | Changes from baseline in NDI at 2nd, 3rd, 4th and 8th week follow-up
Depression scores on Beck's Depression Inventory | Changes from baseline in BDI at 4th and 8th week follow-up
Quality of Life scores on EQ-5D | Changes from baseline in EQ-5D at 2nd, 3rd, 4th and 8th week follow-up
Quality of Life scores on SF-36 | Changes from baseline in SF-36 at 4th and 8th week follow-up
Visual Analogue Scale for pain intensity | Changes from baseline in VAS at 1st, 2nd, 3rd, 4th and 8th week follow-up
Safety profile | At every visit, up to 2 months
  Any adverse events must be documented and reported.
Credibility test | Changes from baseline in credibility test at 4th week follow-up

OTHER OUTCOMES:
Skin Roll Test | Changes from baseline in skinfold thickness and pressure algometer scores at 4th and 8th week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kwan Seo, PhD., KMD, Principal Investigator — Kyunghee University
Locations (1):
- Spine Center, Kyung Hee University Hospital at Gangdong, Seoul, South Korea

REFERENCES:
- [Derived] Seo BK, Lee JH, Kim PK, Baek YH, Jo DJ, Lee S. Bee venom acupuncture, NSAIDs or combined treatment for chronic neck pain: study protocol for a randomized, assessor-blind trial. Trials. 2014 Apr 21;15:132. doi: 10.1186/1745-6215-15-132. PMID 24746224